CLINICAL TRIAL: NCT06081946
Title: Investigation of the Effects of Sleep Provocations on Itch and Pain Sensitivity
Brief Title: Investigation of the Effects of Sleep Fragmentation on Itch and Pain Sensitivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Assistant Professor, Aalborg University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20230028
Record Dates: First submitted 2023-10-02; First posted 2023-10-13 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Histamine; Cowhage; Sleep Fragmentation
MeSH Terms: conditions — Sleep Deprivation | interventions — Histamine

STUDY DESIGN:
Intervention Model Description: The participants will be instructed to wake up at three designated timepoints for three consecutive nights at home.
Masking Description: Participant will be blinded about application of pruritogens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sleep fragmentation (Experimental): This subproject will be conducted in two sessions separated by three nights of sleep fragmentation. Each session will last approximately 2 hours. At the beginning of the first visit and after the last visit, 9 ml of blood will be drawn, and plasma will be isolated. After plasma isolation, the CRP concentration will be analyzed. In each forearm of the participant, a 4x4 cm area will be selected as Area of Interest (AOI). In these selected areas, itch will be induced in both sessions using histamine and cowhage and several tests will be conducted.
  Interventions: Other: Histamine; Other: Cowhage

INTERVENTIONS:
Other: Histamine — Histaminergic itch will be evoked by a 1% histamine solution. A droplet of histamine solution will be placed on the predetermined area on the forearm, and the SPT lancet will be pierced through the histamine with 120 g of pressure for 1-2 seconds
Other: Cowhage — 25 spicules will be inserted in the centre of the predefined skin area on the mandibular area. The spicules will be gently rubbed for 15-20 seconds in circular motion to facilitate epidermal penetration

SUMMARY:
In This experiment, the investigators would like to test following hypotheses regarding the influence of sleep fragmentation on itch:

* To investigate similarity and differences between itch and pain by comparing the effect of sleep deprivation in them.
* To evaluate the inflammatory state induced by sleep fragmentation via the analysis of C-reactive protein (CRP) levels from blood samples.
* To correlate the anxiety and depression scores (evaluated through questionnaires) with itch and pain sensitivity and evaluate how they are affected by sleep fragmentation.

DETAILED DESCRIPTION:
Chronic itch affects approximately a fifth of the global population and is associated with substantial negative consequences for the affected individuals. Furthermore, there is a lack of efficient treatment options for chronic itch.

Poor sleep is a common companion of itch and is often reported by patients with chronic itch. Poor sleep is often characterized by nightly awakenings and troubles falling asleep. This is a significant problem as poor sleep in general is associated with lowered quality of life. While previous research has already established the negative impact of itch on sleep, it is yet to be studied whether the opposite tendency might be true as well. Knowledge about patients with chronic pain has shown that poor sleep can increase the sensitivity to pain and inflammation, and this tendency can also be observed in healthy participants after experimental sleep provocations.

Therefore, the investigators wish to investigate how sleep provocations affect markers of itch in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English
* Access to a smartphone during the experimental nights

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other drugs
* Previous or current history of neurological, dermatological, immunological musculoskeletal, cardiac disorder or mental illnesses (psychiatric diagnosis) that may affect the results (e.g., neuropathy, muscular pain in the upper extremities, anxiety, depression, schizophrenia etc.)
* Moles, wounds, scars, or tattoos in the area to be treated or tested
* Current use of medications that may affect the trial such as antihistamines and pain killers.
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain and itch
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical studies)
* Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of itch | Day 1: 1 minute after every itch inductions
  Immediately following the itch provocations, participants will be instructed to rate the itch intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no itch' and 100 'worst itch imaginable'.
Assessment of itch | Day 2: 1 minute after every itch inductions
  Immediately following the itch provocations, participants will be instructed to rate the itch intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no itch' and 100 'worst itch imaginable'.
Assessment of pain | Day 1: 1 minute after every itch inductions
  Immediately following the itch provocations, participants will be instructed to rate the pain intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no pain' and 100 'worst pain imaginable'.
Assessment of pain | Day 2: 1 minute after every itch inductions
  Immediately following the itch provocations, participants will be instructed to rate the pain intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no pain' and 100 'worst pain imaginable'.

SECONDARY OUTCOMES:
Microvascular reactivity | Day 1: 10 minutes after every itch inductions
  The evoked cutaneous inflammation (quantified by superficial blood perfusion) will be measured by full-field laser perfusion imaging.
Microvascular reactivity | Day 2: 10 minutes after every itch inductions
  The evoked cutaneous inflammation (quantified by superficial blood perfusion) will be measured by full-field laser perfusion imaging.
Touch Pleasantness (TP) | Day 1: 10 minutes after every itch inductions
  Pleasant touch sensation measured using a standardized sensory brush (SENSELab Brush-05, Somedic AB, Hörby, Sweden) exerting a force of 200 to 400 mN. The stimulation consists of three strokes (2 cm in length) over the treated/control areas. The strokes will be applied perpendicularly to the skin and the subject will rate the sensation induced by the brush on a NRS scale labeled "very unpleasant" and "very pleasant" at the extremity and "neutral" at the center.
Touch Pleasantness (TP) | Day 2: 10 minutes after every itch inductions
  Pleasant touch sensation measured using a standardized sensory brush (SENSELab Brush-05, Somedic AB, Hörby, Sweden) exerting a force of 200 to 400 mN. The stimulation consists of three strokes (2 cm in length) over the treated/control areas. The strokes will be applied perpendicularly to the skin and the subject will rate the sensation induced by the brush on a NRS scale labeled "very unpleasant" and "very pleasant" at the extremity and "neutral" at the center.
Mechanically evoked itch (MEI), intensity approach | Day 1: 10 minutes after every itch inductions
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force). This stimulator is moved in intervals of 0.5 cm outside the area of itch provocation.
Mechanically evoked itch (MEI), intensity approach | Day 2: 10 minutes after every itch inductions
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force). This stimulator is moved in intervals of 0.5 cm outside the area of itch provocation.
Mechanically evoked itch, spatial approach | Day 1: 10 minutes after every itch inductions
  The von-Frey filament that better evokes the itch sensation during the assessment of mechanically evoked itch as well as a template of soft plastic are used to map the area of hyperkinesis in the test areas (forearms)
Mechanically evoked itch, spatial approach | Day 2: 10 minutes after every itch inductions
  The von-Frey filament that better evokes the itch sensation during the assessment of mechanically evoked itch as well as a template of soft plastic are used to map the area of hyperkinesis in the test areas (forearms)
Mechanical Pain Thresholds (MPT) | Day 1: 10 minutes after every itch inductions
  This test is conducted using a pinprick set (Aalborg University, Aalborg). The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Thresholds (MPT) | Day 2: 10 minutes after every itch inductions
  This test is conducted using a pinprick set (Aalborg University, Aalborg). The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Sensitivity (MPS), intensity approach | Day 1: 10 minutes after every itch inductions
  This test is conducted with the same pinprick set used to test the MPT. Starting with the lightest, each stimulator is applied at a rate of 2 s on, 2 s off in an ascending order, and the subject will be asked to give a pain rating for each stimulus on a scale from 0-10 (where 0 indicates ''no pain'', and 10 indicates the ''worst imaginable pain'').
Mechanical Pain Sensitivity (MPS), intensity approach | Day 2: 10 minutes after every itch inductions
  This test is conducted with the same pinprick set used to test the MPT. Starting with the lightest, each stimulator is applied at a rate of 2 s on, 2 s off in an ascending order, and the subject will be asked to give a pain rating for each stimulus on a scale from 0-10 (where 0 indicates ''no pain'', and 10 indicates the ''worst imaginable pain'').
Cold Detection Thresholds (CDT) and heat (HPT) detection | Day 1: 10 minutes after every itch inductions
  Thermal cold and heat stimuli will be applied by a contact heat-evoked potential stimulator (PATHWAYS; Medoc Ltd, Ramat Yishai, Israel), placed 5 cm distal to the elbow on the right dorsal forearm
Cold Detection Thresholds (CDT) and heat (HPT) detection | Day 2: 10 minutes after every itch inductions
  Thermal cold and heat stimuli will be applied by a contact heat-evoked potential stimulator (PATHWAYS; Medoc Ltd, Ramat Yishai, Israel), placed 5 cm distal to the elbow on the right dorsal forearm
Cold Detection Thresholds (CDT) and heat (HPT) pain thresholds | Day 1: 10 minutes after every itch inductions
  Thermal cold and heat stimuli will be applied by a contact heat-evoked potential stimulator (PATHWAYS; Medoc Ltd, Ramat Yishai, Israel), placed 5 cm distal to the elbow on the right dorsal forearm
Cold Detection Thresholds (CDT) and heat (HPT) pain thresholds | Day 2: 10 minutes after every itch inductions
  Thermal cold and heat stimuli will be applied by a contact heat-evoked potential stimulator (PATHWAYS; Medoc Ltd, Ramat Yishai, Israel), placed 5 cm distal to the elbow on the right dorsal forearm
Pain to Supra-threshold Heat Stimuli (STHS) | Day 1: 10 minutes after every itch inductions
  The tests will be conducted by using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. The subjects will rate the pain to three suprathreshold heat pain stimuli (starting and ending at 32°C with an increase and decrease of 5°C and 3 s plateau at 50°C).
Pain to Supra-threshold Heat Stimuli (STHS) | Day 2: 10 minutes after every itch inductions
  The tests will be conducted by using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. The subjects will rate the pain to three suprathreshold heat pain stimuli (starting and ending at 32°C with an increase and decrease of 5°C and 3 s plateau at 50°C).
Deep-tissue Pain Sensitivity Measurements | Day 1: 10 minutes after every itch inductions
  Deep-tissue pain sensitivity will be evaluated by cuff pressure stimuli using a computer-controlled cuff algometer (Cortex Technology and Aalborg University, Denmark) including a 13-cm wide tourniquet cuff (VBM, Sulz, Germany) and an electronic visual analog scale (VAS) (Aalborg University, Denmark) for recording of the pain intensity.
Deep-tissue Pain Sensitivity Measurements | Day 2: 10 minutes after every itch inductions
  Deep-tissue pain sensitivity will be evaluated by cuff pressure stimuli using a computer-controlled cuff algometer (Cortex Technology and Aalborg University, Denmark) including a 13-cm wide tourniquet cuff (VBM, Sulz, Germany) and an electronic visual analog scale (VAS) (Aalborg University, Denmark) for recording of the pain intensity.
Pressure Detection and Tolerance Threshold | Day 1: 10 minutes after every itch inductions
  The pressure will be increased by 1 kPa/s and the subject will be instructed to rate the pain intensity continuously on the electronic VAS until the tolerance level is reached.
Pressure Detection and Tolerance Threshold | Day 2: 10 minutes after every itch inductions
  The pressure will be increased by 1 kPa/s and the subject will be instructed to rate the pain intensity continuously on the electronic VAS until the tolerance level is reached.
Temporal Summation of Pain - TSP | Day 1: 10 minutes after every itch inductions
  A total of 10 repeated mechanical pressure stimuli at the PTT level will be delivered at 0.5 Hz (1 s stimulus duration and 1 s interval between stimuli) to the lower leg. A constant pressure of 5 kPa will be applied between the individual pressure stimuli to avoid movement of the cuff. During the 10 repeated stimuli, the subject will continuously rate the pain intensity on a 10 cm continuous VAS.
Temporal Summation of Pain - TSP | Day 2: 10 minutes after every itch inductions
  A total of 10 repeated mechanical pressure stimuli at the PTT level will be delivered at 0.5 Hz (1 s stimulus duration and 1 s interval between stimuli) to the lower leg. A constant pressure of 5 kPa will be applied between the individual pressure stimuli to avoid movement of the cuff. During the 10 repeated stimuli, the subject will continuously rate the pain intensity on a 10 cm continuous VAS.
Conditioned Pain Modulation - CPM | Day 1: 10 minutes after every itch inductions
  The concept of CPM is that a tonic painful stimulus (conditioning stimulus) will inhibit pain evoked simultaneously from another site (test stimulus). The painful conditioned stimulus will be applied simultaneously with the assessment stimulus. The conditioned stimulus will be terminated right after the subject presses the stop button. CPM will be defined as the difference between stimulus during and before the conditioned pain (i.e., "during" minus "before").
Conditioned Pain Modulation - CPM | Day 2: 10 minutes after every itch inductions
  The concept of CPM is that a tonic painful stimulus (conditioning stimulus) will inhibit pain evoked simultaneously from another site (test stimulus). The painful conditioned stimulus will be applied simultaneously with the assessment stimulus. The conditioned stimulus will be terminated right after the subject presses the stop button. CPM will be defined as the difference between stimulus during and before the conditioned pain (i.e., "during" minus "before").
The Itch Catastrophizing Scale | Day 1
  The itch catastrophizing scale is a modified version of the pain catastrophizing scale (PCS), which is a validated questionnaire measuring pain-related thoughts and feelings. The questionnaire consists of 13 items measuring itch-related thoughts and feelings. Each item is rated on a 4-point scale ranging from zero to four, corresponding to thinking/feeling that way during itch 'not at all' and 'very much', respectively.
The Itch Catastrophizing Scale | Day 2
  The itch catastrophizing scale is a modified version of the pain catastrophizing scale (PCS), which is a validated questionnaire measuring pain-related thoughts and feelings. The questionnaire consists of 13 items measuring itch-related thoughts and feelings. Each item is rated on a 4-point scale ranging from zero to four, corresponding to thinking/feeling that way during itch 'not at all' and 'very much', respectively.
The Pittsburg Sleep Quality Index (PSQI) | Day 1
  The PSQI consists of 19 items generating seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The seven component scores can be summarized in a global score ranging from zero to 21 with higher scores reflecting a worse overall quality of sleep.
The Pittsburg Sleep Quality Index (PSQI) | Day 2
  The PSQI consists of 19 items generating seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The seven component scores can be summarized in a global score ranging from zero to 21 with higher scores reflecting a worse overall quality of sleep.
The Hospital Anxiety and Depression Scale (HADS) | Day 1
  The HADS consists of 14 items with two 7-item subscales measuring anxiety and depression symptoms, respectively. Each item is scored on a 4-point scale with zero to three with each subscale ranging from zero to 21. Within both subscales, the scoring is grouped into either normal (0-7), borderline abnormal (8-10), and abnormal (11-21).
The Hospital Anxiety and Depression Scale (HADS) | Day 2
  The HADS consists of 14 items with two 7-item subscales measuring anxiety and depression symptoms, respectively. Each item is scored on a 4-point scale with zero to three with each subscale ranging from zero to 21. Within both subscales, the scoring is grouped into either normal (0-7), borderline abnormal (8-10), and abnormal (11-21).
Positive and Negative Affective Schedule | Day 1
  This 20-item instrument is a psychometric self-report test to assess affect (10 items for positive affect and 10 items for negative affect) and validated for the use in adolescents and adults.
Positive and Negative Affective Schedule | Day 2
  This 20-item instrument is a psychometric self-report test to assess affect (10 items for positive affect and 10 items for negative affect) and validated for the use in adolescents and adults.
Blood Sampling for C-Reactive Protein Analysis | Day 1
  Whole blood samples will be collected from the antecubital vein using a vacutainer blood collection device (S-Monovette, Sarstedt) with a 21-gauge needle.
Blood Sampling for C-Reactive Protein Analysis | Day 2
  Whole blood samples will be collected from the antecubital vein using a vacutainer blood collection device (S-Monovette, Sarstedt) with a 21-gauge needle.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No